CLINICAL TRIAL: NCT03902366
Title: HCV and Co-morbid Alcohol Use Disorders: A Translational Investigation of Antiviral Therapy Outcomes on CNS Function
Status: Completed | Type: Observational
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: Oregon Health and Science University (Other); Portland VA Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: NURA-007-17F; 03967 (Other Grant/Funding Number: Portland VA Medical Center)
Record Dates: First submitted 2019-03-18; First posted 2019-04-04 (Actual); Results first posted 2025-03-27 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Hepatitis C; Alcohol Use Disorder
Keywords: Hepatitis C; Direct-acting antiviral therapies; DAA; Chronic HCV infection; Alcohol Use Disorder
MeSH Terms: conditions — Hepatitis C; Alcoholism | interventions — Neuroimaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood specimens are collected from human subjects by study personnel or the VA phlebotomy lab specifically for research purposes. Research staff centrifuges the blood samples so that components [e.g., plasma, peripheral blood mononuclear cells (PBMCs)] can be collected, frozen, cryopreserved, and contributed to the VA Liver Disease Repository (Director: Dr. Lissi Hansen).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- AUD+/HCV+: * With current Alcohol Use Disorder and with HCV
  * About to initiate DAA therapy for HCV
  Interventions: Diagnostic Test: Neuropsychological assessment; Behavioral: Neuroimaging
- AUD-/HCV+: * Without current Alcohol Use Disorder and with HCV
  * About to initiate DAA therapy for HCV
  Interventions: Diagnostic Test: Neuropsychological assessment; Behavioral: Neuroimaging
- AUD+/HCV-: -With Alcohol Use Disorder and without HCV
  Interventions: Diagnostic Test: Neuropsychological assessment; Behavioral: Neuroimaging
- AUD-/HCV-: -Without Alcohol Use Disorder and without HCV
  Interventions: Diagnostic Test: Neuropsychological assessment; Behavioral: Neuroimaging

INTERVENTIONS:
Diagnostic Test: Neuropsychological assessment — Clinical research staff will complete a standardized neuropsychiatric study visit protocol with eligible participants who provide informed consent. The protocol will be conducted twice for each participant (baseline and 6 months later).
Behavioral: Neuroimaging — Subjects, well characterized with respect to their substance use, will be evaluated with functional magnetic resonance imaging (fMRI) tasks, resting state MRI (rsMRI), high resolution anatomical MRI, standard diffusion weighted imaging (DWI) and high angular resolution diffusion imaging (HARDI) at baseline and 6 months later.

SUMMARY:
The primary objective of this research project is to compare neuropsychiatric functioning, cortical activity, white matter integrity, and immune response among Veterans with and without alcohol use disorder (AUD), before and after direct-acting antiviral (DAA) therapy [a new treatment for chronic infection with the hepatitis C virus (HCV)]. Demographically-matched comparison groups of Veterans without HCV (HCV-, with and without AUD) will similarly be evaluated to determine the relative contribution of HCV and an HCV "cure" to outcomes putatively affected by alcohol abuse.

Two specific aims are proposed.

Aim 1: Determine the impact of DAA therapy and a sustained viral response on central nervous system (CNS) function.

Aim 2: Evaluate the effects of AUD and unhealthy alcohol drinking on DAA therapy outcomes and CNS function.

The information learned will address a critical gap in knowledge concerning the effects of alcohol use on DAA therapy outcomes and will help inform treatment guidelines that could be translated to clinical practice, such as targeted interventions to treat AUD in conjunction with HCV infection and follow-up strategies for patients who successfully complete DAA therapy but then need care for other potential CNS-related outcomes.

DETAILED DESCRIPTION:
Aim 1 will evaluate the impact of DAA therapy on CNS function in Veterans with HCV and will test the hypotheses that following DAA therapy and obtaining a sustained viral response (SVR) [i.e., when the virus continues to be undetectable in blood 12 weeks (or more) after completing therapy], participants will show: i) improved neuropsychiatric outcomes (e.g., cognitive function, fatigue, mood), as compared to baseline (pre-DAA therapy), ii) restored functional connectivity and structural integrity within white matter tracks that had been observed at baseline, and iii) reduced immune activation profiles (e.g., decreased expression of inflammatory biomarkers and restored T cell balance), as compared to baseline. Aim 2 will determine the impact of an active AUD on the neuropsychiatric, neuroimaging, and immunological outcomes observed in aim 1. Participants will be evaluated at two time points [i.e., baseline and 12 weeks post-therapy (week 24)]. Evaluations will incorporate brain imaging methods [i.e., resting state magnetic resonance imaging (MRI), functional MRI, and diffusion tensor imaging] along with clinical and laboratory methods to assess the interactive effects of alcohol use and HCV on brain function. Clinical and laboratory data will include: i) demographic and medical information, ii) neuropsychological measures of attention, memory, and executive function, iii) neuropsychiatric symptom questionnaires (e.g., depression and anxiety), iv) urine and oral fluid collection for medical laboratory tests, and v) blood sample collection for planned experiments (e.g., flow cytometry, quantitative polymerase chain reaction (qPCR), and multiplex immunoassays) and for contribution to the VA Liver Disease Repository.

Evidence-based guidelines for the new DAA therapies are needed (e.g., How much alcohol is too much?). The VA is at the forefront of treating HCV and is now offering DAA therapy to all Veterans with HCV treated within VA health care systems. The proposed studies will address a critical gap in our knowledge concerning the effects of co-morbid HCV and AUD on antiviral therapy outcomes, particularly CNS function and neuropsychiatric symptoms that contribute to addiction and relapse.

ELIGIBILITY:
Inclusion Criteria:

* Adult Veteran (>21 years)
* Able to provide informed consent.

Exclusion Criteria:

* Current substance use disorder other than alcohol (except nicotine or caffeine)
* Medical conditions likely to impact immunological function or central nervous system function (such as HIV, cancer, lupus, stroke, neurodegenerative disease, hepatic encephalopathy, multiple sclerosis, or a traumatic brain injury)
* Visible intoxication or impaired capacity to understand study risks and benefits or otherwise provide informed consent
* Past or present schizophrenia, schizoaffective disorder, or current psychosis or mania
* Visual or auditory impairments that would prevent valid neuropsychiatric testing
* Contraindications to MRI (such as surgical aneurysm clips, pacemaker, prosthetic heart valve, neuro-stimulator, implanted pumps, cochlear implants, metal rods, plates or screws, previous surgery, hearing aids, history of welding, metal shrapnel)

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult Veterans (> 21 years old) who are about to initiate DAA therapy for HCV are recruited into two demographically matched (i.e., similar in terms of age, gender, race, and years of education) groups (n = 30/group): 1) adults with current alcohol use disorder (AUD+/HCV+) and 2) adults without current AUDs (AUD-/HCV+). Two additional groups of demographically-matched adults: 1) without AUD or HCV (AUD-/HCV-) (n = 30), and 2) with AUD and no HCV (AUD+/HCV-) will be recruited as a comparison groups to determine the relative contribution of a history of HCV infection to alcohol-induced brain pathology.
Sampling Method: Non-Probability Sample
Enrollment: 63 (Actual)
Dates: Start 2019-05-16 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2023-12-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer M Loftis, MA PhD, Principal Investigator — VA Portland Health Care System, Portland, OR
Locations (1):
- VA Portland Health Care System, Portland, OR, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of 119 assessed for eligibility, 63 met inclusion criteria (38 AUD-/HCV-, 20 AUD+/HCV-, 5 HCVc) and were enrolled in the study. 17 participants were excluded after enrollment. Due to low recruitment numbers and no significant differences between the HCV groups, individuals with a history of HCV were assigned to one group (HCVc).
Groups:
- Control (AUD-/HCV-): -Without Alcohol Use Disorder and without HCV
  Neuropsychological assessment: Clinical research staff will complete a standardized neuropsychiatric study visit protocol with eligible participants who provide informed consent. The protocol will be conducted twice for each participant (baseline and 6 months later).
  Neuroimaging: Subjects, well characterized with respect to their substance use, will be evaluated with fMRI tasks, rsMRI, high resolution anatomical MRI, standard DWI and high angular resolution diffusion imaging (HARDI) at baseline and 6 months later.
- Alcohol Use Disorder (AUD+/HCV-): -With Alcohol Use Disorder and without HCV
  Neuropsychological assessment: Clinical research staff will complete a standardized neuropsychiatric study visit protocol with eligible participants who provide informed consent. The protocol will be conducted twice for each participant (baseline and 6 months later).
  Neuroimaging: Subjects, well characterized with respect to their substance use, will be evaluated with fMRI tasks, rsMRI, high resolution anatomical MRI, standard DWI and high angular resolution diffusion imaging (HARDI) at baseline and 6 months later.
- HCVc: -Adults with cleared HCV (i.e. no longer test positive for HCV) after receiving treatment (HCVc)
  Neuropsychological assessment: Clinical research staff will complete a standardized neuropsychiatric study visit protocol with eligible participants who provide informed consent. The protocol will be conducted twice for each participant (baseline and 6 months later).
  Neuroimaging: Subjects, well characterized with respect to their substance use, will be evaluated with fMRI tasks, rsMRI, high resolution anatomical MRI, standard DWI and high angular resolution diffusion imaging (HARDI) at baseline and 6 months later.
Period: Baseline
Arm/Group | Control (AUD-/HCV-) | Alcohol Use Disorder (AUD+/HCV-) | HCVc
Started | 27 | 14 | 5
Completed | 27 | 14 | 5
Not Completed | 0 | 0 | 0
Period: Follow-up
Arm/Group | Control (AUD-/HCV-) | Alcohol Use Disorder (AUD+/HCV-) | HCVc
Started | 27 | 14 | 5
Completed | 27 | 14 | 5
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Control (AUD-): -Without Alcohol Use Disorder and without HCV
  Neuropsychological assessment: Clinical research staff will complete a standardized neuropsychiatric study visit protocol with eligible participants who provide informed consent. The protocol will be conducted twice for each participant (baseline and 6 months later).
  Neuroimaging: Subjects, well characterized with respect to their substance use, will be evaluated with fMRI tasks, rsMRI, high resolution anatomical MRI, standard DWI and high angular resolution diffusion imaging (HARDI) at baseline and 6 months later.
- Alcohol Use Disorder (AUD+): -With Alcohol Use Disorder and without HCV
  Neuropsychological assessment: Clinical research staff will complete a standardized neuropsychiatric study visit protocol with eligible participants who provide informed consent. The protocol will be conducted twice for each participant (baseline and 6 months later).
  Neuroimaging: Subjects, well characterized with respect to their substance use, will be evaluated with fMRI tasks, rsMRI, high resolution anatomical MRI, standard DWI and high angular resolution diffusion imaging (HARDI) at baseline and 6 months later.
- HCVc: -Adults treated for HCV
  Neuropsychological assessment: Clinical research staff will complete a standardized neuropsychiatric study visit protocol with eligible participants who provide informed consent. The protocol will be conducted twice for each participant (baseline and 6 months later).
  Neuroimaging: Subjects, well characterized with respect to their substance use, will be evaluated with fMRI tasks, rsMRI, high resolution anatomical MRI, standard DWI and high angular resolution diffusion imaging (HARDI) at baseline and 6 months later.
- Total: Total of all reporting groups
Arm/Group | Control (AUD-) | Alcohol Use Disorder (AUD+) | HCVc | Total
Number analyzed (Participants) | 27 | 14 | 5 | 46
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.70 (14.87) | 59.71 (13.84) | 63.40 (5.37) | 56.59 (14.10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 4 | 1 | 14
  Male | 18 | 10 | 4 | 32
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 0 | 0 | 3
  Not Hispanic or Latino | 24 | 14 | 5 | 43
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 1 | 3
  Asian | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 5 | 2 | 1 | 8
  White | 16 | 12 | 3 | 31
  More than one race | 3 | 0 | 0 | 3
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 27 | 14 | 5 | 46

OUTCOME MEASURES:

1. Primary Outcome: Changes in Neuropsychological Assessment Battery (NAB) Attention Module Scores
Description: The Attention Module is a marker of attentional capacity, working memory, and processing speed. T-scores are derived by converting raw scores using normative tables that account for age and education. T-scores range from 20 to 80 with a mean of 50 and standard deviation of 10. Lower T-scores (below 40) indicate below average performance and higher T-scores (above 60) indicate above-average performance. NAB Attention Module subtests include: Dots, Numbers and Letters, Driving Scenes, Digits Forward, and Digits Backward. Subtest scores were averaged to compute a total score. Change was calculated as the value at 6 months minus the value at baseline. Larger numbers represent greater improvement in attention performance, a score of 0 indicates no change in performance and negative numbers indicate a worsening of attention performance over time.
Time Frame: Baseline and 6 months
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Control (AUD-) | Alcohol Use Disorder (AUD+) | HCVc
Number analyzed (Participants) | 27 | 14 | 5
Units on a scale | 10.99 (3.37) | 0.31 (1.18) | 6.35 (5.92)

2. Primary Outcome: Changes in Neuropsychological Assessment Battery (NAB) Memory Module Scores
Description: The Memory Module is a marker of learning, recall, and recognition memory. T-scores are derived by converting raw scores using normative tables that account for age and education. T-scores range from 20 to 80 with a mean of 50 and standard deviation of 10. Lower T-scores (below 40) indicate below average performance and higher T-scores (above 60) indicate above-average performance. NAB Memory Module subtests include: List Learning, Shape Learning, Story Learning, and Daily Living Memory. Subtest scores were averaged to compute a total score. Change was calculated as the value at 6 months minus the value at baseline. Larger numbers represent greater improvement in memory performance, a score of 0 indicates no change in performance and negative numbers indicate a worsening of memory performance over time.
Time Frame: Baseline and 6 months
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Control (AUD-) | Alcohol Use Disorder (AUD+) | HCVc
Number analyzed (Participants) | 27 | 14 | 5
Units on a scale | 9.07 (1.12) | 1.95 (1.52) | 3.50 (0.71)

3. Primary Outcome: Changes in Neuropsychological Assessment Battery (NAB) Executive Functions Module Scores
Description: The Executive Functions Module of the NAB is a marker of executive function, including problem-solving and mental flexibility. T-scores are derived by converting raw scores using normative tables that account for age and education. T-scores range from 20 to 80 with a mean of 50 and standard deviation of 10. Lower T-scores (below 40) indicate below average performance and higher T-scores (above 60) indicate above-average performance. NAB Executive Function Module subtests include: Mazes, Judgement, Categories, and Word Generation. Subtest scores were averaged to compute a total score. Change was calculated as the value at 6 months minus the value at baseline. Larger numbers represent greater improvement in executive function performance, a score of 0 indicates no change in performance and negative numbers indicate a worsening of executive functioning performance over time.
Time Frame: Baseline and 6 months
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Control (AUD-) | Alcohol Use Disorder (AUD+) | HCVc
Number analyzed (Participants) | 27 | 14 | 5
Units on a scale | 10.65 (0.25) | 5.46 (1.01) | 18.00 (14.14)

4. Primary Outcome: Changes in Alcohol Use Measured Using the Timeline Follow Back (TLFB)
Description: This outcome measure evaluates the change in the number of days of alcohol use from baseline to a 6-month follow-up, using the 30-Day Timeline Followback (TLFB) method. The TLFB is a structured, retrospective interview technique that allows participants to accurately recall their alcohol consumption patterns over the previous 30 days. For this outcome, the number of days on which alcohol was consumed will be assessed at baseline (the start of the study) and again at the 6-month follow-up assessment. A positive change would indicate an increase in the number of days of alcohol use, while a negative change would indicate a reduction in the number of days of alcohol use over the 6-month period.
Time Frame: Baseline and 6 months
Measure: Mean (Standard Deviation); unit: change in the number of days of alcohol
Arm/Group | Control (AUD-) | Alcohol Use Disorder (AUD+) | HCVc
Number analyzed (Participants) | 27 | 14 | 5
change in the number of days of alcohol | 3.78 (9.69) | 44.00 (81.85) | -6.25 (12.5)

5. Primary Outcome: Change in Behavior as Assessed by the Balloon Analogue Risk Task (BART)
Description: The BART is a computerized measure of risk-taking behavior that concurrently measures several domains (i.e., risky decision-making, reward/negative outcome processing) during fMRI scanning.
  The ratio of balloon pumps made to maximum pumps allowed is a measure of risk-taking behavior. A ratio of 1 indicates that a participant inflated the balloon to its maximum allowed pumps, while a ratio closer to 0 suggests that the participant was much more conservative in their approach. Change was calculated as the value at 6 months minus the value at baseline and ranges from -1 to 1. A positive change indicates an increase in risk-taking behavior and a negative change indicates a decrease in risk-taking behavior over time.
Time Frame: Baseline and 6 months
Population: Only 28 of the 46 participants that completed the study, completed both imaging sessions (baseline and 6 months) and were considered for further imaging analyses. Of the 28 participants, one control participant and one participant with cleared HCV (HCVc) were not included in the analysis because task data from at least one timepoint was not collected.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Control (AUD-) | Alcohol Use Disorder (AUD+) | HCVc
Number analyzed (Participants) | 14 | 9 | 3
ratio | -0.018 (0.093) | -0.005 (0.079) | -0.014 (0.164)

6. Primary Outcome: Change in Behavior as Assessed by the Monetary Incentive Delay (MID) Task
Description: The MID is a validated task to examine anticipatory brain responses to reward during fMRI scanning.
  This outcome measure evaluates the change in reaction time (RT) of participants in response to monetary reward cues during the MID. Reaction time is defined as the duration (in milliseconds) from the presentation of the cue to the participant's response (e.g., button press). The MID involves various reward conditions, including different monetary values and probabilities, allowing for an evaluation of participants' anticipatory responses to potential rewards. A positive difference indicates an increase in RT at 6-months compared to baseline, suggesting potential decreases in motivation, cognitive load, or changes in reward sensitivity. Conversely, a negative difference indicates a decrease in reaction time, which may reflect improved motivation, enhanced cognitive processing speed, or increased responsiveness to monetary incentives over time.
Time Frame: Baseline and 6 months
Population: Only 28 of the 46 participants that completed the study, completed both imaging sessions (baseline and 6 months) and were considered for further imaging analyses. Of the 28 participants, two participants (1 HCVc, 1 AUD) were excluded from the study for having incomplete task data.
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Control (AUD-) | Alcohol Use Disorder (AUD+) | HCVc
Number analyzed (Participants) | 15 | 8 | 3
milliseconds | -0.39 (22.83) | 12.77 (19.78) | 3.63 (14.17)

7. Primary Outcome: Change in Fatigue Severity Scale (FSS) Score
Description: The Fatigue Severity Scale (FSS) is a 9-item self-report questionnaire designed to measure level of fatigue. The FSS is graded on a 7-point Likert-like scale ranging from 1 ("strongly disagree") to 7 ("strongly agree"). The score for all 9 items is summed to constitute the FSS score. The minimum FSS score is 7 and the maximum score possible is 63. A higher score represents greater fatigue severity. Change was calculated as the value at 6 months minus the value at baseline and reported here. A higher positive score indicates an increase in fatigue symptoms at 6 months compared to baseline, a lower negative score would indicate a decrease in fatigue symptoms over 6 months and a score of 0 would indicate no change in fatigue symptoms over 6 months.
Time Frame: Baseline and 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control (AUD-) | Alcohol Use Disorder (AUD+) | HCVc
Number analyzed (Participants) | 27 | 14 | 5
score on a scale | 4.87 (12.95) | 2.46 (15.05) | 4.80 (11.97)

8. Primary Outcome: Change in Beck Depression Inventory Second Edition (BDI-II) Score
Description: The Beck Depression Inventory Second Edition (BDI-II) is a 21-question multiple-choice self-report inventory that measures depression. There is a four-point scale for each item ranging from 0-3. The total score can range from 0 to 63 points. Higher scores reflect a great level of depression severity.
Time Frame: Baseline and 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control (AUD-) | Alcohol Use Disorder (AUD+) | HCVc
Number analyzed (Participants) | 27 | 14 | 5
score on a scale | 2.48 (5.98) | 1.92 (7.39) | -0.60 (4.83)

9. Primary Outcome: Change in Fractional Anisotropy (FA) in White Matter Tracts
Description: MRI-based diffusion tensor imaging (DTI) tractography is used to measure fractional anisotropy (FA), an indicator of CNS microstructural integrity. Increases in FA may reflect enhanced fiber organization or myelination, while decreases often indicate demyelination, axonal loss, or reduced coherence of white matter tracts.
  The JHU white-matter tractography atlas was used to extract FA values from 20 structures. Percent change was calculated. A positive number indicates an increase in FA after 6 months and a negative number indicates a decrease in FA from baseline to 6 months.
Time Frame: Baseline and 6 months
Population: Only 28 of the 46 participants that completed the study, completed both imaging sessions (baseline and 6 months) and were considered for further imaging analyses. Of the 28 participants, 4 participants (1 Control, 1 AUD, and 2 HCVc) were not included in the analysis because they had missing or corrupted imaging files.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Control (AUD-) | Alcohol Use Disorder (AUD+) | HCVc
Number analyzed (Participants) | 14 | 8 | 2
percent change
  Left Anterior thalamic radiation | 0.416 (1.791) | -0.612 (2.045) | -1.953 (0.888)
  Right Anterior thalamic radiation | 0.297 (2.158) | -0.768 (1.850) | -1.189 (1.125)
  Left Cingulum cingulate gyrus | 0.341 (2.384) | -0.231 (2.410) | -2.038 (0.731)
  Right Cingulum cingulate gyrus | 0.340 (1.557) | -0.095 (2.210) | -1.218 (0.224)
  Left Cingulum hippocampus | 1.168 (3.190) | 0.259 (2.576) | -2.062 (0.461)
  Right Cingulum hippocampus | -0.113 (1.969) | -0.612 (2.508) | -2.015 (3.444)
  Left Corticospinal tract | 0.337 (1.045) | -0.522 (1.402) | -1.271 (0.737)
  Right Corticospinal tract | 0.130 (1.320) | -0.166 (1.641) | -2.396 (0.712)
  Forceps major | 0.400 (2.038) | -0.295 (2.426) | -2.476 (0.821)
  Forceps minor | 0.317 (3.400) | -0.805 (2.628) | -0.986 (1.692)
  Left Inferior fronto-occipital fasciculus | 0.542 (2.558) | 0.005 (2.503) | -1.700 (0.534)
  Right Inferior fronto-occipital fasciculus | 0.014 (2.693) | -0.410 (1.772) | -1.756 (0.072)
  Left Inferior longitudinal fasciculus | 0.474 (1.764) | -0.002 (1.995) | -1.790 (0.358)
  Right Inferior longitudinal fasciculus | 0.017 (1.971) | -0.234 (1.834) | -2.245 (1.131)
  Left Superior longitudinal fasciculus | 0.424 (1.429) | -0.027 (1.492) | -1.035 (0.744)
  Right Superior longitudinal fasciculus | -0.284 (1.760) | -0.548 (1.260) | -1.840 (0.379)
  Left Superior longitudinal fasciculus, temporal part | 0.540 (1.543) | -0.158 (1.484) | -1.363 (0.398)
  Right Superior longitudinal fasciculus, temporal part | -0.017 (1.474) | -0.671 (1.173) | -1.525 (0.144)
  Left Uncinate fasciculus | 0.462 (3.711) | 0.341 (3.566) | -1.277 (0.614)
  Right Uncinate fasciculus | -0.409 (3.708) | -1.324 (2.321) | -1.609 (1.299)

10. Primary Outcome: Change in Mean Diffusivity (MD) in White Matter Tracts
Description: MRI-based diffusion tensor imaging (DTI) tractography is used to measure mean diffusivity (MD), which is the average rate of water diffusion in all directions within brain tissue. An increase in MD often indicates microstructural disruption, such as axonal loss, demyelination, or increased extracellular space due to edema or atrophy and decreases in MD can reflect cellular proliferation or restricted diffusion, as seen in certain types of gliosis or inflammatory conditions.
  The JHU white-matter tractography atlas was used to extract MD values from 20 structures. Percent change was calculated. A positive number indicates an increase in MD after 6 months and a negative number indicates a decrease in MD from baseline to 6 months.
Time Frame: Baseline and 6 months
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Control (AUD-) | Alcohol Use Disorder (AUD+) | HCVc
Number analyzed (Participants) | 14 | 8 | 2
percent change
  Left Anterior thalamic radiation | -0.740 (1.039) | 0.490 (1.129) | 0.159 (1.507)
  Right Anterior thalamic radiation | -0.827 (0.993) | 0.358 (1.662) | 0.393 (1.856)
  Left Cingulum cingulate gyrus | -0.835 (1.458) | 0.453 (1.269) | -0.288 (1.983)
  Right Cingulum cingulate gyrus | -0.919 (1.566) | -0.177 (2.080) | 0.521 (0.847)
  Left Cingulum hippocampus | -0.932 (2.626) | 0.099 (3.176) | 2.535 (1.258)
  Right Cingulum hippocampus | -0.797 (1.660) | 0.015 (2.180) | 1.131 (4.550)
  Left Corticospinal tract | -0.372 (0.985) | 0.811 (1.180) | 0.522 (0.881)
  Right Corticospinal tract | -0.359 (0.701) | 0.029 (0.928) | 1.169 (1.674)
  Forceps major | -0.474 (1.542) | 0.756 (1.905) | 1.771 (0.407)
  Forceps minor | -0.832 (1.471) | 0.302 (2.164) | -0.674 (1.426)
  Left Inferior fronto-occipital fasciculus | -1.191 (1.161) | -0.014 (1.291) | 0.240 (0.238)
  Right Inferior fronto-occipital fasciculus | -0.862 (1.155) | 0.276 (1.685) | 0.861 (1.655)
  Left Inferior longitudinal fasciculus | -1.128 (1.374) | 0.325 (1.185) | 1.089 (0.099)
  Right Inferior longitudinal fasciculus | -1.006 (1.231) | 0.082 (1.670) | 1.095 (0.914)
  Left Superior longitudinal fasciculus | -0.806 (1.237) | 0.293 (1.154) | 0.249 (0.342)
  Right Superior longitudinal fasciculus | -0.615 (1.116) | 0.276 (1.532) | 0.724 (1.051)
  Left Superior longitudinal fasciculus, temporal part | -0.892 (1.243) | 0.370 (1.109) | 0.516 (0.272)
  Right Superior longitudinal fasciculus, temporal part | -0.777 (1.093) | 0.284 (1.340) | 0.282 (0.952)
  Left Uncinate fasciculus | -1.367 (1.541) | -0.334 (1.792) | -0.633 (0.121)
  Right Uncinate fasciculus | -0.864 (1.716) | 0.582 (2.398) | 0.586 (1.752)

11. Primary Outcome: Changes in Inflammatory Profile Markers: Neutrophil to Lymphocyte Ratio (NLR) and Monocyte to Lymphocyte Ratio (MLR)
Description: Change was calculated as the value at 6 months minus the value and baseline. A positive number indicates an increase in inflammatory markers in plasma samples and a negative value indicates a decrease in inflammatory markers at 6 months.
Time Frame: Baseline and 6 months
Measure: Mean (Standard Deviation); unit: cell count x 10^3/uL [ratio]
Arm/Group | Control (AUD-) | Alcohol Use Disorder (AUD+) | HCVc
Number analyzed (Participants) | 27 | 14 | 5
cell count x 10^3/uL [ratio]
  NLR | -0.36 (0.58) | 0.17 (0.52) | -0.50 (0.42)
  MLR | -0.03 (0.07) | 0.03 (0.07) | 0.45 (0.70)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Control (AUD-) | Alcohol Use Disorder (AUD+) | HCVc
All-Cause Mortality (participants affected / at risk) | 0/27 | 0/14 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/14 | 0/5
Other Adverse Events (participants affected / at risk) | 0/27 | 0/14 | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan: Study Protocol and Statistical Analysis Plan (2024-10-31): https://cdn.clinicaltrials.gov/large-docs/66/NCT03902366/Prot_SAP_000.pdf